CLINICAL TRIAL: NCT04216784
Title: Comparison of Diuretic Effect With Furosemide Alone Versus the Combination of Furosemide and Albumin in Cirrhotic Patients
Brief Title: Compare the Diuretic Effect With Furosemide vs Furosemide and Albumin Combined in Cirrhotic Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study halted prematurely due to staffing.
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19092507-IRB01
Record Dates: First submitted 2019-12-23; First posted 2020-01-03 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Cirrhosis, Liver; Volume Overload; Fluid Overload
MeSH Terms: conditions — Liver Cirrhosis; Edema | interventions — Furosemide; Serum Albumin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Furosemide (Lasix) alone (Active Comparator): Cohort 1 will receive furosemide (Lasix) 40 to 80 mg IVP BID for at least 48 hours
  Interventions: Drug: Furosemide Injection
- Combination of furosemide (Lasix) and albumin (Active Comparator): Cohort 2 will receive combination of furosemide (Lasix) 40 to 80 mg IVP BID and albumin (25%) 12.5 grams IV BID for at least 48 hours
  Interventions: Drug: Furosemide Injection; Drug: Albumin Human

INTERVENTIONS:
Drug: Furosemide Injection — Patient will receive furosemide intravenously
Drug: Albumin Human — Patient will receive albumin (25%) 12.5 gm intravenously
  Arms: Combination of furosemide (Lasix) and albumin

SUMMARY:
A common complication of the progression of cirrhosis is fluid retention (ascites, edema, or pleural effusion). Loop diuretics are the treatment of choice for fluid retention in cirrhotic patients; however, many of these patients demonstrate diuretic resistance, requiring higher doses of the diuretics to achieve adequate diuresis. The cause of this diuretic resistance is hypothesized to be secondary to hypoalbuminemia which has led some providers to give human albumin in combination with loop diuretics to increase intravascular volume and facilitate diuresis. However, this practice remains controversial because minimal data exists to support its efficacy. The purpose of this study is to compare the efficacy of diuretics alone versus diuretics in combination with albumin in cirrhotic patients presenting with fluid retention.

DETAILED DESCRIPTION:
The purpose of this single center, prospective study is to compare the efficacy of two strategies for diuresis in patients with cirrhosis, the use of furosemide (Lasix®) alone versus the combination of furosemide (Lasix ®) and albumin (25%). The investigators will perform a single-center, prospective study with data collected as result of standard of care at Rush University Medical Center (RUMC). Patients who are 18 years of age and older, have diagnosed cirrhosis, and present to RUMC with fluid retention will be identified by the Hepatology and/or Surgery attending and be screened for inclusion in the study. Each patient will be randomized into one of the two cohorts and will have 50% chance of being placed into either cohort. Cohort 1 will receive furosemide (Lasix) 40 to 80 mg intravenous push (IVP) twice a day (BID) for at least 48 hours and cohort 2 will receive combination of furosemide (Lasix) 40 to 80 mg IVP BID and albumin (25%) 12.5 grams BID for at least 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >18 years old)
* Diagnosis of cirrhosis
* Presents with fluid retention as defined as ascites, edema, or pulmonary effusions requiring diuresis.

Exclusion Criteria:

* Patients who are younger than 18 years of age
* Patients who are currently pregnant
* Patients who present with a serum creatinine greater than 2 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lance Lance Lineberger, PharmD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Furosemide (Lasix) Alone | Combination of Furosemide (Lasix) and Albumin
Started | 10 | 11
Completed | 0 | 0
Not Completed | 10 | 11

BASELINE CHARACTERISTICS:
Population: Data was not collected for this study. Study was terminated early due to IRB halting study inclusion and data collection due to drug cost (albumin) funding. Ultimately this dispute resulted in study termination. At no point before the study was halted was data collected on patients enrolled into the study, nor is data going to be collected in patients that were enrolled into the study. Study was anticipated to be prospective randomization for inclusion with data being collected retrospectively
Groups:
- Total: Total of all reporting groups
Arm/Group | Furosemide (Lasix) Alone | Combination of Furosemide (Lasix) and Albumin | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Change in weight defined as weight loss of 1 kilogram
Time Frame: 2-7 days
Population: Data was not collected for this study. Study was terminated early due to IRB halting study inclusion and data collection due to drug cost (albumin) funding. Ultimately this dispute resulted in study termination. At no point before the study was halted was data collected on patients enrolled into the study, nor is data going to be collected in patients that were enrolled into the study.
Arm/Group | Furosemide (Lasix) Alone | Combination of Furosemide (Lasix) and Albumin
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Amount of Urine
Description: The amount of urine produced over 24 hours.
Time Frame: 2-7 days
Population: Data were not reported or collected. At no point before the study was halted was data collected on patients enrolled into the study, nor is data going to be collected in patients that were enrolled into the study.
Arm/Group | Furosemide (Lasix) Alone | Combination of Furosemide (Lasix) and Albumin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Serum Creatinine
Description: Changes in renal function were observed in patients from the two study arms
  . Study was terminated early due to IRB halting study inclusion and data collection due to drug cost (albumin) funding. At no point before the study was halted was data collected on patients enrolled into the study, nor is data going to be collected in patients that were enrolled into the study.
Time Frame: Through completion of study, up to an average of 1 year
Population: Study was terminated early due to IRB halting study inclusion and data collection due to drug cost (albumin) funding. At no point before the study was halted was data collected on patients enrolled into the study, nor is data going to be collected in patients that were enrolled into the study.
Groups:
- Furosemide Alone: patient only received diuretic alone
- Furosemide + Albumin: Patient received furosemide and albumin
Arm/Group | Furosemide Alone | Furosemide + Albumin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Hospital Length of Stay
Description: duration of hospital admission
  Data was not collected for this study. Study was terminated early due to IRB halting study inclusion and data collection due to drug cost (albumin) funding. Ultimately this dispute resulted in study termination. At no point before the study was halted was data collected on patients enrolled into the study, nor is data going to be collected in patients that were enrolled into the study.
Time Frame: Through completion of study, up to an average of 1 year
Population: as for outcome 1
Arm/Group | Furosemide Alone | Furosemide + Albumin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: 30-day Readmission Rates
Description: Number of occurrences that the patient is readmitted after discharge within 30 days
  Data was not collected for this study. Study was terminated early due to IRB halting study inclusion and data collection due to drug cost (albumin) funding. Ultimately this dispute resulted in study termination. At no point before the study was halted was data collected on patients enrolled into the study, nor is data going to be collected in patients that were enrolled into the study.
Time Frame: 30 days from discharge
Population: as for outcome 1
Arm/Group | Furosemide Alone | Furosemide + Albumin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Patient Survival
Description: Patient survival rates to be closely monitored in patients from the two study arms
  Data was not collected for this study. Study was terminated early due to IRB halting study inclusion and data collection due to drug cost (albumin) funding. Ultimately this dispute resulted in study termination. At no point before the study was halted was data collected on patients enrolled into the study, nor is data going to be collected in patients that were enrolled into the study.
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | Furosemide (Lasix) Alone | Combination of Furosemide (Lasix) and Albumin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Study terminated due to IRB halting study inclusion and data collection due to drug cost (albumin) funding. Resulting in study termination."0" denotes that patient data was not collected. Data not collected due to study termination early due to IRB halting study. At no point was data on patients enrolled into the study, nor is data going to be collected in patients that were enrolled. Study was anticipated to be prospective randomization for inclusion with data being collected retrospectively
Description: Study terminated due to IRB halting study inclusion and data collection due to drug cost (albumin) funding. Resulting in study termination."0" denotes that patient data was not collected. Data not collected due to study termination early due to IRB halting study. At no point was data on patients enrolled into the study, nor is data going to be collected in patients that were enrolled. Study was anticipated to be prospective randomization for inclusion with data being collected retrospectively
Arm/Group | Furosemide (Lasix) Alone | Combination of Furosemide (Lasix) and Albumin
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/84/NCT04216784/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT04216784/ICF_001.pdf